CLINICAL TRIAL: NCT07014774
Title: Efficacy of Laser Acupuncture on Carpal Tunnel Syndrome Following Hand Flexor Tendon Repair
Acronym: LASER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Adel Abdel-Hakim Amin, Principle Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mahmoud-005745; Internal2025-Tendon (Other: Internal Use)
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Laser Acupuncture; Flexor Tendon Repair; Hand Surgery; Carpal Tunnel Syndrome (CTS)
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser acupuncture (Experimental): This group includes 30 patients who have had flexor tendon repair surgery and will receive laser acupuncture inform of acupuncture points associated with the median nerve pathway in addition to traditional physical therapy. Patients will receive 3 sessions per week for 8 weeks; each laser acupuncture session lasts 12 minutes, laser applied directly to 12 acupuncture points each point 60 seconds.
  Interventions: Device: Laser acupuncture; Other: Traditional Therapy
- Traditional therapy (Active Comparator): This group includes 30 patients who have had flexor tendon repair surgery and will receive standard postoperative care including physical therapy and medical treatment as needed. Patients will receive 3 sessions per week for 8 weeks; the time of session is 30 minutes according to patient ability.
  Interventions: Other: Traditional Therapy

INTERVENTIONS:
Device: Laser acupuncture — Laser acupuncture is a modern, non-invasive approach to acupuncture that uses low-level laser therapy (LLLT) instead of traditional needles to stimulate acupuncture points. This technique combines the principles of traditional Chinese medicine with modern technology to provide pain relief and promote healing (Chon et al., 2019).
  * Device: UNIPHY PHYACTION 740, made in EEC device.
  * Laser type: Gallium aluminum arsenide laser.
  * Wavelength: 808 nm.
  * Power Output: 200 mW.
  * Dose/energy density: 4J/point.
  * Frequency of treatment: Three times weekly for 8 weeks.
  * Duration: 12 min.
  * Cumulative dose: 48J/point.
  * Target Acupuncture Points: Key points for CTS: PC4 (Ximen), PC6 (Neiguan), PC7 (Daling), PC8 (Laogong), LI4 (Hegu), LI10 (Shousanli), LI11 (Quchi), HT-2 (Qingling), HT7 (Shenmen), HT-8 (Shaofu), LU9 (Taiyuan) and LU10 (Yuji)
  Arms: Laser acupuncture
Other: Traditional Therapy — * Splinting/Bracing: Patients in the two groups will advised to wear a static wrist splint locked at 0_ wrist flexion for at least 8 h at night throughout the entire length of the study as the primary management which reduce pressure on the median nerve.
  * Physical Therapy: Engaging in specific exercises, such as nerve glide exercises and wrist stretches, can improve mobility and reduce symptoms. These exercises aim to restore normal movement of the median nerve and alleviate compression

SUMMARY:
The purpose of this study is to determine the efficacy of laser acupuncture in alleviating CTS symptoms following flexor tendon repair in the hand.

DETAILED DESCRIPTION:
This study holds significant importance for clinical practice, patient care, and research.

* Clinical Practice: It provides a potential framework for physical therapists to design targeted and effective interventions for laser acupuncture on CTS following flexor tendon repair in the hand.
* Patient Care: Improved rehabilitation outcomes can enhance patients' physical functionality, independence, and overall quality of life, addressing a critical gap in post-operative complications.
* Research Advancement: By contributing to the limited body of literature on laser acupuncture in this context, the study can stimulate further research and innovation in carpal tunnel syndrome following hand flexor tendon repair.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20-40 years who have undergone flexor tendon repair surgery.
* Patients who have undergone primary or secondary repair of flexor tendons in the hand at zone 4 (zone of carpal tunnel as it often be complicated by postoperative adhesions due to close quarters and synovial sheath of the carpal tunnel) (Fulchignoni C et al., 2020).
* Surgery occurred within a specific timeframe, often within 6-12 weeks prior to inclusion (Peters SE, Jha B, Ross M., 2021).
* Patient have clinical and electro diagnostic evidence of CTS.
* All patients enrolled to the study will have their informed consent.

Exclusion Criteria:

* Pre-existing neurological disorders.
* Systemic illnesses affecting nerve function (e.g., diabetes).
* Contraindications to laser therapy.
* Pregnancy or breastfeeding.
* Active infections or open wounds in the hand or wrist.
* Previous history of carpal tunnel release surgery or received an injection of steroid for CTS.
* Previous history of brachial plexus injury or median nerve injury.
* Other severe neurological or musculoskeletal conditions.
* Epilepsy or any psychological disorders.
* Cancer.
* Spots over the treated points.
* Pacemaker or implanted devices.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Symptom Relief: | At baseline and after 8 weeks
  Measured by the Visual Analog Scale (VAS) for pain, numbness, and tingling.

SECONDARY OUTCOMES:
- Grip Strength: | Measured at baseline and at the end of the intervention (8 weeks).
  Measured with a hand dynamometer to assess the strength of hand muscles.
- Nerve Conduction Velocity (NCV): | baseline and 8 weeks.
  Measured to assess median nerve conduction before and after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Learning Hospitals Al Kaser Al Ayni Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No